CLINICAL TRIAL: NCT06084520
Title: Translation and Validation of the COMM and ASI-SR - Instruments for Assessing Substance Use Disorder Development in a Swedish Population of Patients With Long-term Pain Treated With Opioids
Brief Title: Translation and Validation of the COMM and ASI-SR
Acronym: COMMISS
Status: Recruiting | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: The Kamprad Family Foundation for Entrepreneurship, Research & Charity (Other)
Responsible Party: Sponsor
Other Study IDs: FoU 2023-00093
Record Dates: First submitted 2023-07-21; First posted 2023-10-16 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Opioid Use; Opioid Use Disorder; Alcohol Use Disorder; Pain, Chronic
MeSH Terms: conditions — Opioid-Related Disorders; Alcoholism; Chronic Pain | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and serum for genetic analysis sampling, but not analysed for the purpose of this study.
  Blood samples for PETH analysis. Dry Blood spott for cannabis analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test group - patients with chronic pain treated with opioids: Patients with long-term, non-cancer-related pain (>3 months) at least 3 days a week, age 18-75 years, who have been treated with opioids for at least 1 month and who can speak, read and write in Swedish, recruited within Uppsala County Primary, Secondary and Tertiary Care.
  Interventions: Diagnostic Test: Current Opioid Misuse Measure (COMM)-SWE; Diagnostic Test: Oral fluid drug test; Diagnostic Test: PETh; Diagnostic Test: ASI-SR; Diagnostic Test: AUDIT; Diagnostic Test: DUDIT; Diagnostic Test: Brief Pain Inventory - BPI; Diagnostic Test: Patient Global Impression of Change PGIC; Diagnostic Test: GAD-7; Diagnostic Test: Patient Health questionnaire (PHQ9); Diagnostic Test: DBS - cannabis test; Other: Sample of Blood for later DNA and immunological analysis in future studies
- Control group - patients with chronic pain not-treated with opioids: Patients with long-term, non-cancer-related pain (>3 months) at least 3 days a week, age 18-75 years, who are not treated with opioids (at inclusion and during the last 3 months) and who can speak, read and write in Swedish, recruited within Uppsala County Primary, Secondary and Tertiary Care.
  Interventions: Diagnostic Test: Oral fluid drug test; Diagnostic Test: PETh; Diagnostic Test: DBS - cannabis test; Other: Sample of Blood for later DNA and immunological analysis in future studies

INTERVENTIONS:
Diagnostic Test: Current Opioid Misuse Measure (COMM)-SWE — Patients in test group should fulfill the the COMM and the battery of validation forms as well as leave the oral fluid for illicit drugs test and whole blod for phosphatidylethanol test.
  Groups: Test group - patients with chronic pain treated with opioids
Diagnostic Test: Oral fluid drug test — Oral fluid sampling to detect drugs. Analysis with LC-HRMS
Diagnostic Test: PETh — Alcohol use detection
  Other Names: Phosphatydilethanol in blood
Diagnostic Test: ASI-SR — Cross-validation form
  Other Names: Addiction Severity Score - Short version
  Groups: Test group - patients with chronic pain treated with opioids
Diagnostic Test: AUDIT — Cross-validation form
  Other Names: Alkohol Use Disorder Identification Test
  Groups: Test group - patients with chronic pain treated with opioids
Diagnostic Test: DUDIT — Cross-validation form
  Other Names: Drug Use Disorder Identification Test
  Groups: Test group - patients with chronic pain treated with opioids
Diagnostic Test: Brief Pain Inventory - BPI — Cross-validation form
  Groups: Test group - patients with chronic pain treated with opioids
Diagnostic Test: Patient Global Impression of Change PGIC — Cross-validation form
  Groups: Test group - patients with chronic pain treated with opioids
Diagnostic Test: GAD-7 — Cross-validation form
  Other Names: Generalized anxiety disorder 7-items scale
  Groups: Test group - patients with chronic pain treated with opioids
Diagnostic Test: Patient Health questionnaire (PHQ9) — Cross-validation form
  Groups: Test group - patients with chronic pain treated with opioids
Diagnostic Test: DBS - cannabis test — cross-validation form
Other: Sample of Blood for later DNA and immunological analysis in future studies — sample collection for future studies

SUMMARY:
The goal of this observational study is to translate the COMM (Current opinion misuse measure) form and validate it using the ASI-SR (Addiction severity score-self report)in a Swedish population of pain patients treated with opioids. The secondary aim is to investigate acceptability of the instrument in a Swedish population of pain patients with long-term opioid treatment (LOT).

The tertiary aim is to investigate the prevalence of alcohol and illicit substance use in a Swedish population of pain patients with LOT.

DETAILED DESCRIPTION:
There is no validated instrument for the assessment of early detection of substance use disorder development in swedish language.

In order to address this gap, investigators plan to translate and validate the COMM questionnaire using the ASI-SR in a Swedish population of pain patients undergoing opioid treatment. In addition, study will investigate the prevalence of illicit substance use in this population and compare it to patients who are not receiving opioid treatment. The collection of material (blood) in the Uppsala Biobank for future analysis of neurobiological processes during long-term pain treatment will be performed.

Phase 1:

Translation of the instrument takes place according to the "Patient-Reported Outcome (PRO) Consortium translation process guidelines"and according to guidelines from the company MAPI ResearchTrust, which owns the rights to use of the instrument.

Phase 2: The subsequent phase entails validating the COMM instrument against the ASI-SR in a Swedish sample of patients experiencing long-term pain, in accordance with the "Cosmin guidelines" [40], and involves the following procedures. Firstly, the reliability of the COMM instrument by examining internal consistency, test-retest consistency, standard error of measurement (SEM), and conducting factor analysis with rotation in a Swedish population of patients with long-term pain andlong-term opioid treatment (LOT)will be assessed. Secondly, validity of the COMM instrument with regard to comprehensiveness, scope, user-friendliness, and predictability within this particular population will be investigated. Furthermore, investigators will assess the acceptability of the instrument among the study population. Finally, exploration of the prevalence of substance use alongside LOT in pain patients and compare it with pain patients who do not receive opioid treatment will be performed. Inclusion goal is to recruit 200 research subjects from various healthcare settings, including primary care, specialized pain care, other specialized care (e.g., Endometriosis Center), and addiction care (addiction medicine program for pain patients) for the test group. Additionally, 200 individuals are planned to be recruited from pain centers and primary care for the control group to measure prevalence rates. The control group will consist of patients with long-term pain who are not undergoing opioid treatment. Since the study involves two groups of patients with long-term pain (with and without opioid treatment), research group will inquire separately if participants are willing to provide blood samples for biomarker analysis of pain (O-link panel) and genetic analysis, which will be stored in the biobank for future research on the effects of opioids.

Validation will be conducted using the results of drug and alcohol analysis from salivatests and blood. Each category, as identified by the original COMMinstrument, will be evaluated against the following instruments:

1. Symptoms and signs of drug abuse (question 1) - AUDIT, DUDIT, ASI-SR, drug and alcohol test
2. Emotional and psychiatric problems (questions 2, 5, 7, 8, 13) - ASI-SR, GAD-7, PHQ9
3. Visitor characteristics/patterns (questions 3, 12, 17) - medical record data
4. Occurrence of untrue statements (doubt/lie/untruth) and drug use (questions 4, 6, 9, 10, 11) - medical record data, drug and alcohol tests
5. Medication use and deviation from prescription (non-compliance) (questions 14, 15, 16) - medical record data, occurrence of overprescription. Pain-related questions will be assessed using the BPI-SF.

In addition, research subjects will also be asked if they would like to be interviewed by a researcher in connection with their consent. Thirty of the initial research subjects who respond positively will undergo a semi-structured interview, where ease of use will be examined using the "think aloud" method. This involves asking subjects about their thoughts on the forms, including their understanding of the questions, language choices, and any possible negative associations. The interviews will then be reviewed using qualitative content analysis.

Moreover, an extensive assessment will be undertaken, involving the input of 10 esteemed professionals in Sweden who specialize in various fields related to this subject matter, such as pain doctors, addiction medicine doctors, psychologists, behavioral scientists, and others. These experts will be approached to provide their valuable insights by responding to a set of carefully devised questions concerning the evaluation of content validity. Their estimations will serve as the fundamental basis for calculating the Content Validity Index (CVI).

In order to collect and analyze the health data, information from medical records, relevant forms, and laboratory responses are compiled into a study database and then transferred to a statistics program. To ensure internal consistency and reliability, Cronbach's alpha is used, with the expectation that it will be higher than 0.70 at a significance level of p<0.05. Additionally, the agreement between the two test occasions of COMM is assessed using the intraclass correlation coefficient (ICC). The ICC is classified as satisfactory if below 0.40, good if between 0.40-0.59, and excellent if between 0.60-0.70. The correlation between the results of COMM and the ASI-SR is examined using both the Pearson and Spearman correlation coefficients, which are calculated for the respective clusters of questions in the form. Furthermore, confirmatory factor analysis with rotation is employed to investigate the relationship between different clusters or dimensions of questions that can be identified for correlation purposes. The discriminant validity of ASI-SR composite scores and external validity measures are determined by calculating the intercorrelation matrix between COMM groups of questions, ASI-SR composite scores, and external validation measures. The minimum requirement for correlation is set at >0.40. Statistical processing is conducted using SPSS, SAP, and Amos programs. It should be noted that the qualitative aspect of the study is not covered by the statistical plan. In terms of prevalence estimation, both the test group and the control group will be described using descriptive statistics. The occurrence of addictive drugs, non-prescribed drugs, and measures of alcohol use (PETh) during the last three weeks in both groups will be compared using a chi-square test. Odds analysis will be performed to assess secondary use of illegal substances, parallel dependence on other substances, and drugs and alcohol during the length of the study.

ELIGIBILITY:
Inclusion Criteria:

Intervention group:

* Patients with long-term, non-cancer-related pain (>3 months) at least 3 days a week
* opioid treatment for at least 1 month during last 6 months
* age 18-75 years
* fluent in spoken and written Swedish.

Control group:

* Patients with long-term, non-cancer-related pain (>3 months) at least 3 days a week
* no opioid treatment at inclusion and during last 3 months
* age 18-75 years
* fluent in spoken and written Swedish

Exclusion Criteria:

* ongoing diseases or conditions that prevents the patient from completing to the study according to the doctor's assessment
* serious cognitive disorder that makes answering the questions impossible. - - ongoing or treated cancer in the last 10 years
* Insufficient knowledge of Swedish

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic pain patients (18-75 years old) within Uppsala County treated both in Primary care, Secondary care ( Endometrios center) and Tertiary care ( Pain and Addiction clinic)
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
COMM - Current opioid misuse version Swedish version | Baseline
  COMM is based on 17 questions, all of which are answered on a 5-point Likert scale.
  As the original COMM instrument has identified 5 categories of questions, each area will be assessed against the following instruments:
  1. Symptoms and signs of drug abuse (question 1) - AUDIT, DUDIT, ASI-SR, drug and alcohol test
  2. Emotional and psychiatric problems (questions 2,5,7,8,13) - ASI-SR, GAD-7, PHQ9
  3. Visitor characteristics/patterns (questions 3,12,17) - medical record data
  4. Occurrence of untrue statement (doubt/lie/untruth) and drug use (questions 4,6,9,10,11) - medical record data, drug and alcohol tests

SECONDARY OUTCOMES:
ASI-SR Addiction severity index - short release | Baseline
  This instrument is based on interview questions that are used for addiction monitoring by calculating "composite scores", mathematical score measures that are sensitive to change and that are used for follow-up and research. The scoring measures are produced according to a standardized model from the National Board of Health and Welfare (2017). Each domain is calculated in point measures.
COMM - 2nd test | 1 week after baseline
  COMM is based on 17 questions, all of which are answered on a 5-point Likert scale. For retest consistency.
AUDIT Alcohol Use Disorder Identification Test | Baseline
  Scoring system, (0-40)where increase of the points reflects increased risk of problematic alcohol use.
BPI-Brief Pain Inventory - short form | Baseline
  BPI-SF measures ongoing intensity and impact of pain on different areas of life (eg activity, sleep, well-being). Questions are answered in scale 0-10. From there you can calculate the indexes "Pain Intensity" and "Pain Interference".
Patient global impression of change - PGI-C | Baseline
  7-grade scale (-3-+3)where the lowest points indicate negative and highest points indicate positive change.
Drug Use Disorder Identification Test (DUDIT) | Baseline
  Scoring system,(0-44) where increase of the points reflects increased probability of drug abuse syndrome.
Patient Health Questionnaire PHQ9 | Baseline
  Depression Assesment scoring system, (0-15) where <4 is no need of depression treatment, and >15 identifies need of pharmacologic or other depression treatment
Drug detection test - saliva | baseline
  Analysis performs with tandem high-resolution liquid mass spectrometry (LC-HRMS) positive/negative results according to the intern cut-off standard
PETh - Phosphatidylethanol in blood | baseline
  Test monitoring alcohol consumtionduring last 3 weeks monitoring. Results talking: no alcohol use < 0.05 microg/l , moderate use 0.05-0.30, regular high. amount use >30microg/l.
Cannabis in DBS ( Dry blood spott) | baseline
  Analysis performs with tandem high-resolution liquid mass spectrometry (LC-HRMS) positive/negative results according to the intern cut-off standard
Generalized anxiety disorder (GAD-7)[ | baseline
  7-items scale, Summary score (0-21), where severity of anxiety increase with more points: <5 no anxiety, 6-10 mild, 11-16 moderate, <17 severe

OTHER OUTCOMES:
Descriptive characteristics of the group | baseline
  Age, sex, level of education, work status is requested in the survey, duration of treatment and pain condition and number of visits to healthcare in the last six months (specifically acute visits), diagnosis for which the preparation is prescribed, preparation and dose and actual amount prescribed in the last 6 months and any signs of overuse or problematic use For evaluating factor structure principal component analyses (PCA) .

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Karlsten, PhD, Principal Investigator — Uppsala University
Locations (1):
- Multidisciplinary Pain Center, Uppsala, Uppland, Sweden

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT06084520/Prot_SAP_000.pdf